CLINICAL TRIAL: NCT04273815
Title: A Phase Ib, Open-label, Dose Escalation and Expansion Study to Evaluate the Tolerance , Pharmacokinetics and Effectiveness of TQ-A3334 Tablets in Patients With Advanced Non-small Cell Lung Cancer
Brief Title: A Study to Evaluate the Tolerance, Pharmacokinetics and Efficacy of TQ-A3334 Tablets
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQA3334-Ⅰ-02
Record Dates: First submitted 2020-02-16; First posted 2020-02-18 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — anlotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQ-A3334 tablets (Experimental): TQ-A3334 tablets administered orally on day1, 8, 15 in 21-day cycle.
  Interventions: Drug: TQ-A3334
- TQ-A3334 tablets + anlotinib capsules (Experimental): TQ-A3334 tablets administered orally on day1, 8, 15 in 21-day cycle plus Anlotinib capsules given orally in fasting conditions , once daily in 21-day cycle (14 days on treatment from Day 1-14, 7 days off treatment from Day 15-21).
  Interventions: Drug: TQ-A3334; Drug: Anlotinib

INTERVENTIONS:
Drug: TQ-A3334 — TQ-A3334 is a highly efficient and highly selective TLR-7 agonist. TLR-7 can induce the release of a series of pro-inflammatory cytokines, including IFN-α (interferon-α), IL-12 (Interleukin 12), TNF-α, and promote the maturation and antigen presentation of dendritic cells, play an antitumor effect.
Drug: Anlotinib — Anlotinib is a multi-target receptor tyrosine kinase inhibitor.
  Arms: TQ-A3334 tablets + anlotinib capsules

SUMMARY:
This is a study to evaluate the tolerance, dose-limiting toxicity (DLT), and maximum tolerated dose (MTD) of single and multiple oral doses of TQ-A3334 and observe the efficacy of TQ-A3334 in combination with anlotinib capsules in patients with non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1.Understood and signed an informed consent form; 2. 18 years old and older; Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 1; life expectancy ≥12 weeks; 3.Histologically confirmed advanced non-small cell lung cancer; 4. Has received at least two systemic chemotherapy regimens which is failure or intolerance; 5. At least one measurable lesion（ based on RECIST1.1）; 6. The main organs function are normally; 7. Male or female subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 6 months after the last dose of study (such as intrauterine devices , contraceptives or condoms) ；No pregnant or breastfeeding women, and a negative pregnancy test are received within 7 days before the randomization; 8. In addition to the above criteria, the extended research phase must meet the following criteria: EGFR and ALK are negative; or patients with positive test results of EGFR and ALK are resistant or intolerant after receiving the targeted drug treatment.

Exclusion Criteria:

* 1. Small cell lung cancer; 2. Other malignant tumors that have appeared or are currently present within 5 years, except for cured cervical carcinoma in situ, non-melanoma skin cancer; 3. Has received chemotherapy, surgery, radiotherapy, the last treatment from the first dose less than 4 weeks, or oral targeted drugs for less than 5 half-lives, or oral fluorouracil pyridine drugs for less than 14 days, mitomycin C and nitrosourea for less than 6 weeks; 4. Expect to use any active vaccine against infectious diseases within 28 days before the first administration or during the study period; 5. Immunosuppressive therapy with immunosuppressive agents or systemic or absorbable local hormones (dosage > 10 mg/day prednisone or other therapeutic hormones) is required for the purpose of immunosuppression, and is still in use for 2 weeks after the first administration; 6. Active autoimmune diseases that require systemic treatment have occurred within 2 years before the first administration; 7. Hypersensitivity to TQB3804 or its excipient; 8. Has uncontrollable symptoms of brain metastases, spinal cord compression, cancerous meningitis; 9. Has unrelieved toxicity reactions ≥ grade 1 due to previous treatment; 10. Imaging (CT or MRI) shows that tumor invades large blood vessels or the boundary with blood vessels is unclear; 11. Has thyroid dysfunction that requires drug treatment within 6 months before the first administration; 12. Has multiple factors affecting oral medication; 13.Has any severe acute complications before the first administration; 14. Have participated in other clinical trials within 4 weeks before the first administration; 15. According to the judgement of the researchers, there are other factors that may lead to the termination of the study; 16. In addition to the above criteria, the extended research phase must meet the following criteria: 1) Pathologically diagnosed as central, hollow lung squamous cell carcinoma, or non-small cell lung cancer with hemoptysis ; 2) EGFR and ALK are positive untreated with relevant targeted drugs; 3) Has received anlotinib hydrochloride capsules.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-07-06 (Actual); Primary Completion 2021-01-31 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AE) | Baseline up to 21 days
  The occurrence of adverse events and serious adverse events.
Dose limited toxicity (DLT) and Maximum tolerable dose (MTD) | Baseline up to 21 days
  DLT defined as any of the following events occurring during the study related to drugs ： （1） ≥grade 3 non-hematologic toxicity; （2）Grade 4 neutropenia, thrombocytopenia, and hemoglobin reduction confirmed by at least 2 tests within 2 days; （3）Grade 3 neutropenia with fever confirmed at least 2 times within 2 days; （4）Immune-related interstitial pneumonia ≥ grade 2 ；. （5）Decreased ventricular ejection fraction ≥ grade 2 ； （6）Retinal vein occlusion (RVO), uveitis ≥ grade 2 ; MTD defined as the highest dose level at which less than or equal to 2 of 6 subjects experience dose limiting toxicity (DLT).

SECONDARY OUTCOMES:
Tmax | 5minutes, 15minutes, 0.5hour, 45minutes, 1hour, 1.5hour, 4hour, 12hour, 24hour, 48hour, 96hour, 144hour after oral administration on day 1 and day 29; 30min before oral administration on day 1, day8, day15,day22 and day 29.
  To characterize the pharmacokinetics of TQ-A3334 by assessment of time to reach maximum plasma concentration.
Cmax | 5minutes, 15minutes, 0.5hour, 45minutes, 1hour, 1.5hour, 4hour, 12hour, 24hour, 48hour, 96hour, 144hour after oral administration on day 1 and day 29; 30min before oral administration on day 1, day8, day15,day22 and day 29.
  Cmax is the maximum plasma concentration of TQ-A3334 or metabolite(s).
t1/2 | 5minutes, 15minutes, 0.5hour, 45minutes, 1hour, 1.5hour, 4hour, 12hour, 24hour, 48hour, 96hour, 144hour after oral administration on day 1 and day 29; 30min before oral administration on day 1, day8, day15,day22 and day 29.
  t1/2 is time it takes for the blood concentration of TQ-A3334 or metabolite(s) to drop by half.
AUC0-t | 5minutes, 15minutes, 0.5hour, 45minutes, 1hour, 1.5hour, 4hour, 12hour, 24hour, 48hour, 96hour, 144hour after oral administration on day 1 and day 29; 30min before oral administration on day 1, day8, day15,day22 and day 29.
  To characterize the pharmacokinetics of TQ-A3334 by assessment of area under the plasma concentration time curve from zero to infinity.
Overall response rate (ORR) | up to 96 weeks
  Percentage of Participants Achieving Complete Response (CR) and Partial Response (PR).
Progression-free survival (PFS) | up to 96 weeks
  PFS defined as the time from randomization until the first documented progressive disease (PD) or death from any cause.
Duration of Response (DOR) | up to 96 weeks
  Time from tumor first assessment to CR or PR to first assessment to PD (Progressive Disease) or death from any cause.
Disease control rate（DCR） | up to 96 weeks
  Percentage of Participants Achieving Complete Response (CR) and Partial Response (PR) and Stable Disease (SD).

CONTACTS AND LOCATIONS:
Locations (1):
- Jinling Hospital, Nanjing, Jiangsu, China